CLINICAL TRIAL: NCT05988294
Title: Pulmonary Function, Respiratory Muscle Strength and Functional Capacity Response to Pilates Exercises in Patients with Inhalation Injury After Thermal Burn.
Brief Title: Pilates Exercises in Patients with Inhalation Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004571
Record Dates: First submitted 2023-07-29; First posted 2023-08-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-08

CONDITIONS: Inhalation Injury
Keywords: Pilates exercises; Pulmonary Function; Respiratory Muscle Strength; Functional Capacity Response; Inhalation Injury; Thermal Burn
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Pilates Group) (Experimental): Participants will receive Pilates exercises for 60 minutes followed by conventional physical therapy program for 45 minutes, 3 days/ week for 12 weeks.
  Interventions: Other: Pilates exercises; Other: Conventional physical therapy exercise program
- Group B (Control Group) (Other): Participants will receive conventional physical therapy program (diaphragmatic deep breathing exercises, bronchial hygiene techniques, assisted cough, stretching exercises and ROM exercises for both upper and lower limbs) for 45 minutes, 3 days/ week for 12 weeks.
  Interventions: Other: Conventional physical therapy exercise program

INTERVENTIONS:
Other: Pilates exercises — One-hour Pilates exercise program was given by a certified trainer to patients three times per week for 12 weeks. The exercise program followed the basic principles of the Pilates method. Our protocol comprised the following components of Pilates-based exercises: strength and stabilization, flexibility and range of motion, proper body alignment, balance, coordination, and body awareness. Resistance bands and 26 cm Pilates balls were used as supportive equipment. The exercise sections consisted of 5 minutes breathing, 10 minutes warm-up, 35 minutes conditioning phase and 10 minutes cool-down.
  Arms: Group A (Pilates Group)
Other: Conventional physical therapy exercise program — Diaphragmatic deep breathing exercises, bronchial hygiene techniques, assisted cough, stretching exercises and ROM exercises for both upper and lower limbs for 45 minutes, 3 days/ week for 12 weeks.

SUMMARY:
Inhalation injury is a composite of multiple insults including: supraglottic thermal injury, subglottic airway and alveolar poisoning, and systemic poisoning from absorbed small molecule toxins. These contaminant insults independently affect each of the pulmonary functions as well as having a direct effect on systemic physiology. Further, anatomic characteristics can predispose patients to inhalation injury. For example, an infant will develop airway obstructions much faster than an adult due to reduced airway diameter. Understanding the contributions of each of these pathologies to the patient's disease is critical to managing inhalation injury.

DETAILED DESCRIPTION:
Extra lung mucus secretions, injured mucosa, contaminants, and aspirated substances should be handled in their early stages. In the case of fibrinous material transudates, compromised mucociliary secretions and mucosal slough must be cleared. There are different methods to assist the clearance of secretions as bronchoscopy, ventilator, mucolytics, suction, and chest physiotherapy.

In Pilates method (PM), several muscles are activated, including the muscles involved in breathing, especially to improve the expiratory function, which remains contracted during the inspiratory and expiratory phase. Breathing control is fundamental during the execution of PM exercises, where the practitioner learns how to breathe properly as an essential part of each exercise through forceful exhaling followed by complete inhaling. Thus, adequate breathing aids in controlling movements, and therefore, the method can be regarded as an indirect strategy for respiratory muscle training. It is known that poor control of breathing can result in compensation and lung volumes and respiratory muscle performance, with several factors involved.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in both sexes and their age will range from 20-50 years.
2. Six weeks after deep second-degree thermal burn with inhalation injury (until complete healing) with 35%-40% total body surface area (TBSA).
3. Patients suffering from retained secretions which did not respond to medical treatment. (4) All patients should be clinically and medically stable.

(5) All patients should have the same medical treatment.

Exclusion Criteria:

1. Participants with a history of regular physical activity (regular exercise habit > 3 times/ week or >150 min/ week) in the last 6 months.
2. Participants with less than an 85% attendance rate at the sessions.
3. Participants with any dysfunction that limit physical activity such as neurological disorders, chronic obstructive pulmonary disease, uncontrolled hypertension, malignancy, cardiovascular diseases, deep vein thrombosis, rheumatoid arthritis, orthopedic problems, such as fracture on the pelvic or limbs, a visual impairment, or hearing impairments and contractures.
4. Smokers.
5. Pregnant females.
6. Obese participants (BMI > 30 kg/m2).
7. Participants use non-invasive mechanical ventilation and intubation or need for intensive clinical support and/or transfer to the Intensive Care Unit.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 12 weeks
  Forced vital capacity (FVC) will be measured by using spirometer
forced expiratory volume in 1 second (FEV1) | 12 weeks
  forced expiratory volume in 1 second (FEV1) will be measured by using spirometer
peak expiratory flow (PEF) | 12 weeks
  peak expiratory flow (PEF) will be measured by using spirometer

SECONDARY OUTCOMES:
Respiratory muscle strength | 12 weeks
  The inspiratory muscle strength will be verified by means of the maximum inspiratory pressure (MIP) and the expiratory muscular strength by means of maximum expiratory pressure (MEP) by using the digital Manovacuometer
Functional capacity | 12 weeks
  By using 6-Minute Walk Test (6-MWT) that measures the maximum distance walked in a period of 6 min to assess the submaximal level of the functional capacity of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Elimy, PhD, Study Director — Lecturer of basic science, Faculty of Physical Therapy Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: Study protocol